CLINICAL TRIAL: NCT04769466
Title: Development of a Reminiscence Therapy Online Platform With Machine Learning to Increase Engagement With People Living With Dementia and Their Care Partners
Brief Title: LifeBio Memory Digital Reminiscence Platform
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benjamin Rose Institute on Aging (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1908-216; 1R44AG069566-01 (NIH)
Record Dates: First submitted 2020-09-28; First posted 2021-02-24 (Actual); Results first posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-08

CONDITIONS: Dementia; Cognitive Impairment
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Staff (Experimental): Staff will be trained in the platform, and complete life story interviews with residents at their facilities. Upon completion of training, staff will complete surveys regarding it's effectiveness and utility, and following the completion of the interview, the resident's life story books, summary materials, and staff tools will be delivered four weeks later. Life story materials are meant to assist staff in providing more personalized care and a mechanism for residents to feel more deeply understood.
  Interventions: Other: LifeBio Memory
- Residents (Experimental): Residents will be screened for their cognitive status and compete interviews with a researcher prior to participation in the life story interview. Residents will then be interviewed again at T3 about four weeks after the life story books, summaries, and staff materials have been delivered.
  Interventions: Other: LifeBio Memory

INTERVENTIONS:
Other: LifeBio Memory — LifeBio Memory is a digital reminiscence therapy platform designed to collect the life stories of older adults to generate personalized life storybooks that capture their unique narratives and social histories. Life story booklets, summaries, and materials are also developed as mechanisms for sharing this story and for staff to provide enhanced person-centered care.

SUMMARY:
Non-pharmacological interventions and person-centered care strategies are important elements of care for people with Alzheimer's disease and related dementias. Life story work, which uses written and oral life histories to elicit conversation and memories, is an effective intervention for individuals with dementia; however, because of the time-consuming nature of generating useful life story materials, has not been widely implemented in nursing homes and other care environments. LifeBio Inc. will develop an easy-to-use reminiscence therapy platform - LifeBio MemoryTM - with a novel machine-learning-based application that converts speech to text and generates life stories to serve as an interactive tool to cultivate communication between people living with dementia and their family and caregivers.

DETAILED DESCRIPTION:
This project offers the unique and timely opportunity to evaluate the feasibility, acceptability, and efficacy of LifeBio Memory's effectiveness as a solution for improving quality of life and quality of care for older adults in long-term care settings, as well as relationships with staff caregivers. This project will implement the the newly developed LifeBio Memory platform and train caregivers in X sites across the state of Ohio, with X residents and X staff participating in a feasibility trial. The program will be evaluated using three waves of data collection from staff during training and throughout implementation, as well as pre-post resident data to evaluate the effectiveness of the new intervention.

The LifeBio Memory platform addresses the need for an intuitive, artificial intelligence-driven solution to the traditionally labor-intensive process of collecting, sharing, and celebrating the life stories of older adults, as well as the development of tools for staff caregivers to enhance person-centered care practices and care-planning. It has great potential for improving psychosocial outcomes for participants, enhancing relationships between care staff and residents, and a cost-effective way to identify ways in which life stories can be used to provide a foundation for preference-based, personalized care.

Residents will be interviewed at baseline, then again at follow-up (4 weeks later), staff members being trained to utilize the LifeBio Memory application and provide feedback on the materials, as well as completed a survey at baseline, again at follow-up

ELIGIBILITY:
Inclusion Criteria (Staff):

* Work within a residential care facility participating in the study
* Speak and read English
* Able to provide own transportation to and from interviews with residents

Inclusion Criteria (Residents

* Must reside within a participating residential care facility
* Must be at least 55 years of Age
* Must speak and read English
* Have a Dementia diagnosis
* Have a Score of at least 15 on the Mini Mental State Examination

Exclusion Criteria (Residents)

* Residents will be excluded from the study if they show signs of rapid cognitive decline or physical deterioration over the last 6 months, as evidence by information gained during screening.

Ages: 18 Years to 112 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Orsulic-Jeras, MA, Principal Investigator — Benjamin Rose Institute on Aging
Locations (1):
- Benjamin Rose Institute on Aging, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Staff | Residents
Started | 71 | 163
Completed | 53 | 107
Not Completed | 18 | 56

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Staff | Residents | Total
Number analyzed (Participants) | 53 | 107 | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 0 | 50
  >=65 years | 3 | 107 | 110
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 49 | 76 | 125
  Male | 3 | 31 | 34
  Unknown or Not Reported | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 46 | 101 | 147
  Unknown or Not Reported | 6 | 6 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 12 | 16
  White | 47 | 91 | 138
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 53 | 107 | 160

OUTCOME MEASURES:

1. Primary Outcome: Change in Center for Epidemiological Studies Depression Scale (CES-D) From Baseline
Description: 10-item Measure of depressive symptomatology; Scale: 0 (rarely or none of the time) to 3 (most or almost all of the time); Possible scores range from 0 (minimum) to 30 (maximum). Higher scores indicate higher frequency of reported depressive symptomology.
Time Frame: Baseline, After intervention (4 weeks from baseline)
Population: Staff were not assessed for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Residents
Number analyzed (Participants) | 107
score on a scale
  Baseline | 7.04 (5.18)
  Post Intervention | 6.09 (5.06)
Statistical Analysis 1: Comparison: Residents; T-Test; Test type: Other; p = 0.020, t-test, 1 sided

2. Primary Outcome: Change in Satisfaction With Care in the Nursing Home Scale From Baseline
Description: Measurement of resident satisfaction with care in a long-term care facility; 8-items measured on a scale of 1 = generally yes and 0 = generally no; Possible scores range from 0 (minimum) to 8 (maximum). Higher scores indicate higher satisfaction with care at the resident's facility.
Time Frame: Baseline; After intervention (4 weeks from baseline)
Population: Staff were not assessed for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Residents
Number analyzed (Participants) | 107
score on a scale
  Baseline | 6.95 (1.42)
  Post Intervention | 6.84 (1.39)
Statistical Analysis 1: Comparison: Residents; T-Test; Test type: Other; p = 0.223, t-test, 1 sided

3. Primary Outcome: Change in Quality of Life Alzheimer's Disease (QoL-AD) From Baseline
Description: 13-item Quality of life scale for an individual living with Alzheimer's Disease: rated on a scale of 1 (poor) to 4 (excellent); Possible scores range from 13 (minimum) to 52 (maximum). Higher scores indicate higher quality of life.
Time Frame: Baseline; After intervention (4 weeks from baseline)
Population: Staff were not assessed for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Residents
Number analyzed (Participants) | 107
score on a scale
  Baseline | 35.60 (6.33)
  Post Intervention | 34.70 (5.34)
Statistical Analysis 1: Comparison: Residents; T-Test; Test type: Other; p = 0.036, t-test, 2 sided

4. Primary Outcome: Change in Cohen-Mansfield Agitation Inventory (CMAI) - Short Form From Baseline
Description: 14-item Measurement of agitation that was completed by the staff for each resident they were assigned to conduct a life story interview with at baseline and post-intervention (proxy completed by staff on behalf of each resident) rated on a scale: 1 (never) to 5 (several times an hour) scores can range from 14-70, with higher scores indicating higher frequency of agitated behaviors of persons living with dementia as reported by those staff conducting their life story interviews.
Time Frame: Baseline; After intervention (4 weeks from baseline)
Population: Staff were not assessed for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Residents
Number analyzed (Participants) | 107
score on a scale
  Baseline | 17.13 (8.41)
  Post Intervention | 16.23 (4.58)
Statistical Analysis 1: Comparison: Residents; Test type: Other; p = 0.131, t-test, 1 sided

5. Primary Outcome: Change in Staff Attitudes Towards Residents Scale From Baseline
Description: Measurement of the attitudes of long term care staff towards the residents under their care includes 4-items on a 5-pt scale of 1= never to 5=always, scores ranging from 4 to 20, higher scores indicate more positive attitudes toward residents.
Time Frame: Baseline; After intervention (4 weeks from baseline)
Population: Residents were not assessed for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Staff
Number analyzed (Participants) | 53
score on a scale
  Baseline | 16.43 (1.87)
  Post Intervention | 16.32 (1.82)
Statistical Analysis 1: Comparison: Staff; Test type: Other; p = 0.351, t-test, 1 sided

6. Primary Outcome: Change in Individualized Care Instrument (ICI) Subscale - Knowing the Person - From Baseline
Description: 13-item subscale of the ICI scale "knowing the person"; rated on a scale from 1 (strongly disagree) to 4 (strongly agree); Possible scores range from 13 (minimum) to 52 (maximum). Higher scores indicate staff feel they know the resident more.
Time Frame: Baseline; After intervention (4 weeks from baseline)
Population: Residents were not assessed for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Staff
Number analyzed (Participants) | 53
score on a scale
  Baseline | 41.09 (5.91)
  Post Intervention | 42.15 (6.64)
Statistical Analysis 1: Comparison: Staff; Test type: Other; p = 0.08, t-test, 1 sided

7. Primary Outcome: Change in The UCLA 3-Item Loneliness Scale From Baseline
Description: 3-item Measurement of feelings of loneliness; rated on a scale: 1 (hardly ever) to 3 (often), ranging from 3 to 9, higher scores indicate higher feelings of loneliness.
Time Frame: Baseline; After intervention (4 weeks from baseline)
Population: Staff were not assessed for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Residents
Number analyzed (Participants) | 107
score on a scale
  Baseline | 4.50 (1.79)
  Post Intervention | 4.46 (1.80)
Statistical Analysis 1: Comparison: Residents; T-Test; Test type: Other; p = 0.400, t-test, 1 sided

8. Primary Outcome: Resident Satisfaction With the LifeBio Memory Program
Description: A total of 9-items were developed from the pilot and current study to understand resident's acceptance and satisfaction with the LifeBio Memory program. Participants answered either "no" (0) or "yes" (1) to each item, with total scores ranging from 0 to 9 (higher scores indicating high satisfaction with the LifeBio Memory program).
Time Frame: After intervention (4 weeks from baseline)
Population: Staff were not assessed for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Residents
Number analyzed (Participants) | 107
score on a scale | 6.42 (2.11)

9. Primary Outcome: Change in Perceived Importance of Life Story Work Among Staff
Description: 3-item measure related to the importance of life story work with residents; items are rated on a scale from 1 = strongly disagree to 5 = strongly agree, scores ranging from 3 to 15, with higher scores indicating staff feeling life story work is more important.
Time Frame: Baseline; After intervention (4 weeks from baseline)
Population: Residents were not assessed for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Staff
Number analyzed (Participants) | 53
score on a scale
  Baseline | 13.32 (1.92)
  Post-Intervention | 12.79 (2.13)
Statistical Analysis 1: Comparison: Staff; Test type: Other; p = 0.011, t-test, 2 sided

10. Primary Outcome: Staff Satisfaction With LifeBio Memory Program
Description: On the follow-up post-evaluations, staff were asked to rate their overall satisfaction with the LifeBio Memory program. A total of 8-items developed from the pilot and current study were rated on a 1 (strongly disagree) to 5 (strongly agree) scale. Possible scores range from 8 (minimum) to 40 (maximum). Higher scores indicate higher satisfaction with the program.
Time Frame: After intervention (4 weeks from baseline)
Population: Residents were not assessed for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Staff
Number analyzed (Participants) | 53
score on a scale | 33.57 (5.00)

11. Primary Outcome: Change in Sense of Competence in Dementia Care Staff (SCIDS) Scale From Baseline
Description: 17-item measurement of staffs' overall sense of dementia care competence; rated on a scale: 1 (not at all) to 4 (very much) with scores potentially ranging from 17-68, higher scores indicating higher sense of competence in dementia care among staff.
Time Frame: Baseline; After intervention (4 weeks from baseline)
Population: Residents were not assessed for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Staff
Number analyzed (Participants) | 53
score on a scale
  Baseline | 55.35 (8.82)
  Post Intervention | 55.48 (10.03)
Statistical Analysis 1: Comparison: Staff; Test type: Other; p = 0.459, t-test, 1 sided

12. Primary Outcome: Change in Person-Centered Care Assessment Tool [Sub-Scales I and II] From Baseline
Description: 10-item measurement of staff experience with person-centered care in their current care community; rated on a scale: 1 (strongly disagree) to 5 (strongly agree), scores ranging from 10-50, higher scores indicating higher agreement with experience providing person-centered care.
Time Frame: Baseline; After intervention (4 weeks from baseline)
Population: Residents were not assessed for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Staff
Number analyzed (Participants) | 53
score on a scale
  Baseline | 39.70 (5.54)
  Post Intervention | 37.96 (6.99)
Statistical Analysis 1: Comparison: Staff; Test type: Other; p = 0.033, t-test, 1 sided

13. Primary Outcome: Change in Direct Care Worker Job Satisfaction Scale From Baseline
Description: 9-item measurement of staff satisfaction with different aspects of their job; rated on a Scale: 1 (very dissatisfied) to 4 (very satisfied), potential scores ranging from 9-36, higher scores indicating higher satisfaction with their job.
Time Frame: Baseline; After intervention (4 weeks from baseline)
Population: Residents were not assessed for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Staff
Number analyzed (Participants) | 53
score on a scale
  Baseline | 27.66 (4.25)
  Post Intervention | 26.85 (5.08)
Statistical Analysis 1: Comparison: Staff; Test type: Other; p = 0.103, t-test, 1 sided

14. Primary Outcome: Change in Individualized Care Instrument (ICI) Subscale - Resident Autonomy Subscale - From Baseline
Description: 15-item Measurement of staff perceptions about resident's autonomy; rated on a Scale: 1 (never) to 5 (very frequently), potential scores ranging from 15-75, higher scores indicating staff perceiving residents having more frequent autonomy.
Time Frame: Baseline; After intervention (4 weeks from baseline)
Population: Residents were not assessed for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Staff
Number analyzed (Participants) | 53
score on a scale
  Baseline | 58.46 (7.78)
  Post Intervention | 58.44 (8.95)
Statistical Analysis 1: Comparison: Staff; Test type: Other; p = 0.494, t-test, 1 sided

15. Primary Outcome: Change in Individualized Care Instrument (ICI) Subscale - Staff and Resident Communication Subscale - From Baseline
Description: 7-item measurement of staff perceptions of their communication with residents; rated on a Scale: 1 (never) to 4 (always), scores ranging from 7-28. higher scores indicating higher frequency of staff to resident communication about their care.
Time Frame: Baseline; After intervention (4 weeks from baseline)
Population: Residents were not assessed for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Staff
Number analyzed (Participants) | 53
score on a scale
  Baseline | 20.72 (3.88)
  Post Intervention | 21.15 (4.03)
Statistical Analysis 1: Comparison: Staff; Test type: Other; p = 0.214, t-test, 1 sided

16. Primary Outcome: Change in Individualized Care Instrument (ICI) Subscale - Staff to Staff Communication Subscale - From Baseline
Description: 10-item measurement of staff perceptions of staff to staff level communication, rated on a scale from 1 (never) to 4 (always), scores ranging from 10-40, higher scores indicating more frequent staff to staff communication.
Time Frame: Baseline; After intervention (4 weeks from baseline)
Population: Residents were not assessed for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Staff
Number analyzed (Participants) | 53
score on a scale
  Baseline | 27.02 (6.85)
  Post Intervention | 26.30 (7.23)
Statistical Analysis 1: Comparison: Staff; Test type: Other; p = 0.199, t-test, 1 sided

17. Primary Outcome: Staff Perceptions About the Feasibility of the LifeBio Memory Program Protocol
Description: 7-items were developed (rated on a 1 = strongly disagree to 5 = strongly agree response scale) and administered on the follow-up post-evaluation to understand staff's perceptions about the feasibility of the program protocol once interviews were complete and materials (i.e., Action Plans, Life Story books, Snapshots) were delivered (e.g., Within the first 2-weeks of delivery, I was able to present the residents' Action Plans during a team meeting"). Possible scores range from 7 (minimum) to 35 (maximum). Higher scores indicate higher feasibility with the implementation of program materials.
Time Frame: After intervention (4 weeks from baseline)
Population: Residents were not assessed for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Staff
Number analyzed (Participants) | 53
score on a scale | 26.26 (5.58)

18. Secondary Outcome: Change in Mini Mental Status Examination (MMSE) From Baseline
Description: Screening for resident cognitive status, scores can range from 0-30, lower scores indicate more cognitive impairment (higher scores indicate less cognitive impairment).
Time Frame: Baseline; After intervention (4 weeks from baseline)
Population: Staff were not assessed for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Residents
Number analyzed (Participants) | 107
score on a scale
  Baseline | 21.07 (3.91)
  Post Intervention | 19.72 (4.80)

19. Secondary Outcome: Change in Staff Adequate Knowledge of Residents' Care Preferences From Baseline
Description: 1-item asked of staff for each resident they interviewed on a scale of 1 = not at all well, to 5 = extremely well ("How well do you know the resident's care preferences?")
Time Frame: Baseline; After intervention (4 weeks from baseline)
Population: This item was filled out by staff per resident they interviewed - therefore it is measured per resident.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Residents
Number analyzed (Participants) | 107
score on a scale
  Baseline | 2.76 (0.90)
  Post-Intervention | 3.54 (0.97)
Statistical Analysis 1: Comparison: Residents; Test type: Other; p < .001, t-test, 2 sided

20. Secondary Outcome: Change in Staff Adequate Knowledge of Residents' Life Stories From Baseline
Description: 1-item asked of staff for each resident they interviewed on a scale of 1 = not at all well, to 5 = extremely well ("How well do you know the resident's life story?")
Time Frame: Baseline; After intervention (4 weeks from baseline)
Population: This item was filled out by staff per resident they interviewed - therefore it is measured per resident.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Residents
Number analyzed (Participants) | 107
score on a scale
  Baseline | 2.68 (0.92)
  Post-Intervention | 3.58 (0.93)
Statistical Analysis 1: Comparison: Residents; Test type: Other; p < .001, t-test, 2 sided

21. Other Pre Specified Outcome: Length of Time Staff Spent on LifeBio Memory Training
Description: Item related to staff time spent on LifeBio Memory training
Time Frame: Training was assigned to be completed within one week of baseline. Staff objective knowledge was measured immediately after completing the training videos.
Population: A total of 71 staff completed the post-training survey. However, 18 staff did not complete the entire study protocol due to various reasons (e.g., time constraints, left facility).
Measure: Count of Participants; unit: Participants
Arm/Group | Staff
Number analyzed (Participants) | 71
Participants
  The length of time you spent on training was appropriate. | 61
  The length of time you spent on training was too long. | 8
  The length of time you spent on training was too short. | 2

22. Other Pre Specified Outcome: Preparedness Of Staff Conducting Life Story Interviews
Description: Staff self-rated preparedness to conduct life story interviews with residents and set up their accounts following training; two 1-item survey questions rated on a scale from 1 = strongly disagree to 6 = strongly agree. Higher score on each item means stronger agreement towards feelings of being prepared to conduct a life story interview with a person living with dementia using the LifeBio Memory app and setting up their account using the LifeBio Memory app.
Time Frame: as for outcome 21
Population: A total of 71 staff completed the post-training survey, however 18 staff did not complete the entire study protocol due to various reasons (e.g., time constraints, left facility).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Staff
Number analyzed (Participants) | 71
score on a scale
  Average feeling of preparedness to conduct the life story interviews using the LifeBio Memory app | 5.04 (0.992)
  Average feeling of preparedness to set up an account using the LifeBio Memory app after training. | 4.92 (1.118)

23. Other Pre Specified Outcome: Staff Training Needs Being Met With LifeBio Memory Training
Description: Staff overall feelings of needs being met with the LifeBio Memory Training Program. Staff were asked, "Overall, how well does the LifeBio Memory App training meet your needs?" On a scale from 1 = not well at all to 5 = extremely well.
Time Frame: as for outcome 21
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Staff
Number analyzed (Participants) | 71
score on a scale | 3.73 (0.916)

24. Other Pre Specified Outcome: Staff Objective Knowledge of LifeBio Memory Training Content
Description: Staff completed an 11-item quiz post-training (tested on content detailed in the training videos). It was a multiple choice type quiz, and average score represents total number of correct items on the quiz. Scores could range from 0 to 11, with the staff ranging from 5-items correct to 11-items answered correctly. Higher scores indicate higher number of quiz items answered correctly.
Time Frame: as for outcome 21
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Staff
Number analyzed (Participants) | 71
score on a scale | 9.37 (1.68)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the date of enrollment in the study to the last date a subject was active in the study. This time frame was approximately a 22-month period.
Description: Not different from clinicaltrials.gov
Arm/Group | Staff | Residents
All-Cause Mortality (participants affected / at risk) | 0/71 | 15/163
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/163
Other Adverse Events (participants affected / at risk) | 0/71 | 0/163

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-05-26): https://cdn.clinicaltrials.gov/large-docs/66/NCT04769466/Prot_SAP_ICF_000.pdf